CLINICAL TRIAL: NCT02865564
Title: Effect of Lactobacillus Reuteri DSM17938 in Neonates Treated With Antibiotics on Emergence of Functional Gastrointestinal Disorders, Body Composition, Mineral Bone Density and Fecal Microbiota in Infancy
Brief Title: Effect of Lactobacillus Reuteri DSM17938 in Neonates Treated With Antibiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Jana Lozar Krivec, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UPKLjubljana
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Diseases; Colic
Keywords: Probiotics; Anti-Bacterial Agents; Infant, Newborn; Gastrointestinal Microbiome; Colic; Gastrointestinal Diseases; Body Composition; Bone Density; Randomized Controlled Trial; Lactobacillus reuteri; Pediatrics; Feces; ultrasonography; High-Throughput Nucleotide Sequencing; Electric Impedance; Surveys and Questionnaires
MeSH Terms: conditions — Gastrointestinal Diseases; Colic | interventions — Ampicillin; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group will receive 5 drops, a minimum of 100 million live Lactobacillus reuteri DSM 17938 a day during antibiotic treatment (empirical treatment for neonatal sepsis with ampicillin and gentamicin) and 6 consecutive weeks after finishing the antibiotic treatment.
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938; Drug: ampicillin and gentamicin
- Placebo group (Placebo Comparator): Placebo group will receive 5 drops of maltodextrin in the some oil suspension a day during antibiotic treatment (empirical treatment for neonatal sepsis with ampicillin and gentamicin) and 6 consecutive weeks after finishing the antibiotic treatment.
  Interventions: Dietary Supplement: Placebo; Drug: ampicillin and gentamicin

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938
  Other Names: BioGaia
  Arms: Intervention group
Dietary Supplement: Placebo
  Arms: Placebo group
Drug: ampicillin and gentamicin

SUMMARY:
The aim of the study is to elucidate the relationship between postnatal antibiotic administration on development of gut microbiota and possible protective influence of simultaneously administration of probiotic during antibiotic therapy on development of gut microbiota, functional gastrointestinal disorders of infancy, weight gain and body composition.

DETAILED DESCRIPTION:
The study is double-blind, placebo-controlled randomised trial and is composed from two parts. First part of the study aims to examine any difference in gut microbiota after postnatal antibiotic administration between the neonates who received probiotic Lactobacillus reuteri DSM 17938 or placebo and to compare the gut microbiota of patients to microbiota of healthy newborns. Second part of the study aims to determine whether probiotic L. reuteri DSM 17938 supplementation to antibiotic therapy has any beneficial influence on incidence of functional gastrointestinal disorders of infancy and body composition and bone density 6 weeks and one year after inclusion in the study.

Additionally the associations of the clinical parameters with the composition and developmental characteristics of fecal microbiota during antibiotic treatment in children will be evaluated; relevant clinical data such as mode of delivery, child's nutrition, health problems, growth and developmental attributes which could be found associated with fecal microbial community, will be tracked and statistically evaluated for the investigated population.

ELIGIBILITY:
Inclusion Criteria:

* term neonates whom antibiotic treatment will be introduced due to clinical suspicion of infection

Exclusion Criteria:

* gestational age under 37 weeks
* birth weight less than 2500 grams
* congenital malformations/syndromes
* perinatal hypoxia
* who had received probiotics before the randomization
* have had cow's milk protein allergy diagnosed during the study
* patient who will be treated with antibiotic for less than 5 days

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Functional gastrointestinal dysfunction | At 6 months of age
  Questionnaire [/]
Composition of gut microbiota in infants - 1 | At 6 weeks after intervention
  [colony-forming units/ml; /]
Infants crying duration time | At 6 months of age
  Questionnaire [/]
Composition of gut microbiota in infants - 2 | At one year of age
  [colony-forming units/ml; /]

SECONDARY OUTCOMES:
Infant weight - 1 | At 6 months of age
  [kg]; to calculate body mass index
Bone mineral density in infants - 1 | At 6 months of age
  Z-score [/]
Infant height - 1 | At 6 months of age
  [m]; to calculate body mass index
Infant weight - 2 | At 12 months of age
  [kg]; to calculate body mass index
Bone mineral density in infants - 2 | At 12 months of age
  Z-score [/]
Infant height - 2 | At 12 months of age
  [m]; to calculate body mass index
Body composition of infants - 1 | At 6 months of age
Body composition of infants - 2 | At 12 months of age

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lozar Krivec J, Bratina P, Valcl A, Lozar Manfreda K, Petrovcic A, Benedik E, Obermajer T, Bogovic Matijasic B, Setina U, Rupnik M, Mahnic A, Paro-Panjan D. Effects of Limosilactobacillus reuteri DSM 17938 in neonates exposed to antibiotics: a randomised controlled trial. Benef Microbes. 2024 Oct 31;16(2):157-169. doi: 10.1163/18762891-bja00049. PMID 39486439